CLINICAL TRIAL: NCT04088032
Title: A Pilot Neoadjuvant Clinical Trial of Combination Therapy With Abemaciclib, Durvalumab (MEDI4736), and an Aromatase Inhibitor in Locally Advanced Hormone Receptor Positive Breast Cancer
Brief Title: Neoadjuvant Study of Abemaciclib, Durvalumab, and an Aromatase Inhibitor Early Stage Breast Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Per sponsor
Sponsor: Alison Stopeck (Other)
Collaborators: Eli Lilly and Company (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Alison Stopeck, Division Chief Hematology/Oncology, Stony Brook University
Organization: Stony Brook University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00174 Neoadj Breast Pilot
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer Female; Locally Advanced Breast Cancer; Hormone Receptor Positive Malignant Neoplasm of Breast
MeSH Terms: interventions — abemaciclib; durvalumab; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): Experimental treatment
  Interventions: Drug: Abemaciclib, durvalumab and aromatase inhibitor

INTERVENTIONS:
Drug: Abemaciclib, durvalumab and aromatase inhibitor — Subjects will receive standard therapy with an aromatase inhibitor (exemestane, anastrozole, or letrozole), combined with the experimental treatment of abemaciclib and durvalumab

SUMMARY:
The purpose of this study is to test the efficacy, safety and tolerability of a combination of immunotherapy and anticancer drugs presurgery in patients with hormone-receptor positive breast cancer.

DETAILED DESCRIPTION:
The primary hypothesis is that a Programmed death-ligand 1 (PD-L1) immune checkpoint inhibitor combined with a Cyclin-dependent kinase 4/6 (CDK4/6) inhibitor will be well tolerated in early stage, hormone receptor positive (HR+) breast cancer patients treated with neoadjuvant endocrine therapy (NET). The secondary hypothesis and biomarker based endpoint is that patients with HR positive locally advanced breast cancer with low to intermediate stromal tumor-infiltrating lymphocytes (TILs) will demonstrate an increase in stromal TILs following NET when combined with abemaciclib and durvalumab for 4 cycles (16 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. A signed, written informed consent will be obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
2. Postmenopausal women age ≥ 18 years at time of study entry. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Women <50 years of age receiving luteinising hormone-releasing hormone (LHRH) agonist for ovarian suppression are also eligible for the study but must initiate LHRH agonist therapy at least 2 weeks prior to starting on study intervention.
   * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
3. Histologically confirmed estrogen and/or progesterone positive invasive breast cancer, defined as either estrogen and/or progesterone receptor (ER/PR) staining >10%, AND Human Epidermal Growth Factor Receptor 2 (HER2) negative by either Immunohistochemistry (IHC) or Fluorescent in situ Hybridization (FISH).
4. Clinical stage II-III disease with no clinical or radiologic evidence of metastatic disease. Patients must have a measurable primary breast lesion as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 guidelines.
5. Eastern Cooperative Oncology Group (ECOG) status < 1.
6. Patient must be able to swallow pills.
7. Adequate organ and marrow function as defined below and in Table 1:

   * Hemoglobin ≥ 9 g/deciliter
   * Absolute neutrophil count ≥ 1,500/mm3
   * Platelet count ≥ 100,000/mm3
   * Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2 × institutional upper limit of normal (ULN)
   * Bilirubin ≤ 1.5 × ULN; for subjects with documented/suspected Gilbert's disease, bilirubin ≤ 2 × ULN
   * Creatinine clearance ≥ 50 mL/min as determined by the Cockcroft-Gault equation, or creatinine ≤1.5 x ULN
8. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
9. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Any serious preexisting medical condition(s) that would place the patient at increased risk for toxicities including interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, history of major surgical resection involving the stomach or small bowel.
2. Body weight < 30 kg (or 66.5 lbs.). If during the study, the patient's weight drops to < 30 Kg (or 66.5 lbs), they will be withdrawn from the study.
3. Females who are pregnant or lactating.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, severe active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement or compromise the ability of the subject to give written informed consent
5. Active or prior documented autoimmune disease within the past 2 years. NOTE: Subjects with vitiligo, Grave's disease, Hashimoto's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are eligible
6. History of significant cardiac disease including heart failure, ventricular arrhythmia, or prolonged QT syndrome.
7. Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or a preexisting chronic condition resulting in baseline ≥ Grade 2 diarrhea.)
8. History of primary immunodeficiency, or subjects who are known to be HIV (Human Immunodeficiency Virus ) positive
9. History of organ transplant that requires use of immunosuppressives
10. Known allergy or reaction to any of the study drugs.
11. Other invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured
12. Major surgical procedure (as defined by the investigator) within 30 days prior to the first dose of study drugs or still recovering from prior surgery
13. Known history of tuberculosis
14. Subjects who are known to be hepatitis B or C positive
15. History of prior therapy with a checkpoint (PD-L1/PD-1) including durvalumab or CDK4/6 inhibitor
16. History of prior ipsilateral radiation therapy to the cancer-affected breast
17. History of prior therapy with an investigational anticancer therapy within 6 weeks prior to the first dose of study drugs
18. Prior chemotherapy or aromatase inhibitor therapy for breast cancer
19. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal, topical, and inhaled corticosteroids or systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
20. Patients who must take strong cytochrome cytochrome P450 (CYP3A) inhibitors such as clarithromycin, diltiazem, verapamil, itraconazole, or ketoconazole
21. Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
22. Concurrent enrollment in another therapeutic clinical study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Through study completion, up to 24 weeks
  The primary endpoints will be safety and tolerability of the study intervention

SECONDARY OUTCOMES:
Pathologic response at surgery | At the time of definitive surgery
  Pathologic response at surgery by Preoperative Endocrine Prognostic Index (PEPI) score
Pathologic response at surgery | At the time of definitive surgery
  Pathologic response at surgery by change in Ki-67% from pre and surgical biopsies

OTHER OUTCOMES:
Change in the number of T cells | At the time of definitive surgery
  Change in subtype of T cell infiltrates and spatial relationship of T cells to tumor cells (number of T cells withing the tumor)
Change in the number of T regs cells | At the time of definitive surgery
  Change in number of T regs per tumor spatial unit
Change in the number of macrophages | At the time of definitive surgery
  Change in number of myeloid derived immunosuppressive cells (M1 vs M2 macrophages) per tumor spatial unit
Changes in immune markers in the tumor specimens and/or peripheral blood | At the time of definitive surgery
  Change in gene expression immune signatures (RNA quantification)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Stopeck, MD, Study Director — Stony Brook University; Lea Baer, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Cancer Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No